CLINICAL TRIAL: NCT05877339
Title: The Effect of Exercise on Fatigue in White-collar Workers
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2023
Record Dates: First submitted 2023-04-09; First posted 2023-05-26 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Exercise; Fatigue
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Fertility

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Osteoartritis: Patients with osteoarthritis among the participants
  Interventions: Diagnostic Test: Survey
- Fibromyalgic Disease: Patients with fibromyalgia among the participants
  Interventions: Diagnostic Test: Survey
- Control Group: Healthy people
  Interventions: Diagnostic Test: Survey

INTERVENTIONS:
Diagnostic Test: Survey — Survey

SUMMARY:
A survey will be conducted on the Internet for desk workers. The questionnaire; International Physical Activity Questionnaire will be filled out to evaluate the exercise level of the participants, the visual analog scale to question the general pain levels, and the fatigue severity questionnaire to investigate the fatigue levels. The patients will also be divided into the presence of osteoarthritis, the presence of fibromyalgia, and healthy group, and an evaluation will be made between the groups.

DETAILED DESCRIPTION:
A survey will be conducted on the Internet for desk workers. The questionnaire; International Physical Activity Questionnaire will be filled out to evaluate the exercise level of the participants, the visual analog scale to question the general pain levels, and the fatigue severity questionnaire to investigate the fatigue levels. The patients will also be divided into the presence of osteoarthritis, the presence of fibromyalgia, and healthy group, and an evaluation will be made between the groups.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years old
* white-collar worker
* agree to participate in the study

Exclusion Criteria:

* history of musculoskeletal surgery
* the presence of illness that will prevent him/her from exercising

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20-75 years old white-collar worker
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Survey | through study completion, an average of 1 month
  The patients were evaluated by completing the International Physical Activity Questionnaire, visual pain scale and fatigue severity scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)